CLINICAL TRIAL: NCT02297815
Title: Comparative Effectiveness of Broad vs. Narrow Spectrum Antibiotics for Acute Respiratory Tract Infections in Children
Brief Title: Comparative Effectiveness of Antibiotics for Respiratory Infections
Acronym: CEARI
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 13-010595
Record Dates: First submitted 2014-11-17; First posted 2014-11-21 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-04

CONDITIONS: Acute Otitis Media; Acute Sinusitis; Group A Streptococcal Pharyngitis
Keywords: antibiotic use; effectiveness; acute respiratory infections; pediatrics
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Broad-spectrum antibiotics: Children diagnosed with an acute respiratory tract infections (ARTI) and prescribed Broad-spectrum antibiotics.
  Interventions: Drug: Broad-spectrum antibiotics
- Narrow-spectrum: Children diagnosed with an acute respiratory tract infections (ARTI) and prescribed Narrow-spectrum antibiotics.
  Interventions: Drug: Narrow-spectrum antibiotics

INTERVENTIONS:
Drug: Broad-spectrum antibiotics — Amoxicillin-clavulanate, azithromycin, cefdinir, cefprozil, cefuroxime axetil, cefadroxil, cephalexin
  Groups: Broad-spectrum antibiotics
Drug: Narrow-spectrum antibiotics — Amoxicillin, Penicillin
  Groups: Narrow-spectrum

SUMMARY:
The purpose of this study is to identify and use patient centered outcomes to compare narrow-spectrum and broad-spectrum antibiotics for the treatment of common acute respiratory tract infections (ARTIs) in children.

DETAILED DESCRIPTION:
Outpatient, ARTIs account for the vast majority of antibiotic exposure to children, and roughly half of these antibiotic prescriptions are inappropriate. Although unnecessary antibiotic prescribing for viral infections has significantly decreased, there has been a substantial increase in prescribing of broad-spectrum antibiotics to treat ARTIs when narrow-spectrum antibiotics are indicated. Primary care providers, patients, and caregivers would benefit from studies assessing the implications of alternate antibiotic regimens for these common infections. Specifically, it remains unclear if treating common ARTIs with broad-spectrum antibiotics leads to an improvement in patient outcomes compared to treatment with narrow-spectrum antibiotics, particularly considering the increasing threat posed by antimicrobial resistance. Because of the lack of large comparative effectiveness studies with patient-centered outcomes addressing this issue, professional guidelines and expert recommendations are conflicting, and, as a result, practice patterns vary considerably. Therefore, using patient-centered outcomes, we aim to compare narrow-spectrum and broad-spectrum antibiotics for the treatment of common ARTIs in children. To accomplish this, we will perform a prospective cohort study of children receiving antibiotics for ARTI across a comprehensive pediatric healthcare network. We will conduct telephone interviews with parent's of children who receive antibiotic treatment for an ARTI. We will assess previously identified patient-centered outcomes included a health-related quality of life measure, occurrence of side effects, missed school/daycare, parent missed commitments and/or required additional childcare and symptoms were still present on day 3 after diagnosis.

ELIGIBILITY:
Inclusion Criteria:

We included children between six months and 12 years old, diagnosed with an ARTI (acute otitis media, acute sinusitis, Group A streptococcal [GAS] pharyngitis) using International Classification of Diseases diagnosis codes and prescribed an antibiotic. For GAS pharyngitis, the child also had a positive rapid streptococcal test.

Exclusion Criteria:

* Diagnosed with multiple ARTIs
* Diagnosed with another non-ARTI bacterial infection
* Prescribe antibiotics in the past 30 days
* Non-English speaking families
* If GAS pharyngitis diagnosis, age < 3 years

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Child diagnosed with an ARTI and prescribed antibiotics during an outpatient visit in the CHOP primary care network.
Sampling Method: Probability Sample
Enrollment: 2472 (Actual)
Dates: Start 2014-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Gerber, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Narrow Spectrum Antibiotic: Children diagnosed with an ARTI and prescribed a narrow-spectrum antibiotic
- Broad-Spectrum Antibiotic: Children diagnosed with an ARTI and prescribed a Broad-spectrum antibiotic
Period: Overall Study
Arm/Group | Narrow Spectrum Antibiotic | Broad-Spectrum Antibiotic
Started | 1604 | 868
5-10 Day Interview | 1604 | 868
14-20 Day Interview | 1368 | 728
Completed | 1368 | 728
Not Completed | 236 | 140
Not completed — Lost to Follow-up | 236 | 140

BASELINE CHARACTERISTICS:
Groups:
- Narrow Spectrum Antibiotics: Child prescribed with the following at time of diagnosis:
  Acute otitis media: Amoxicillin Acute sinusitis: Amoxicillin Streptococcal pharyngitis: Penicillin or Amoxicillin
- Non-narrow Spectrum Antibiotics: Child prescribed with the following at time of diagnosis:
  Acute otitis media: Amoxicillin-Clavulanate, Azithromycin, Cefdinir, Cefprozil, Cefuroxime Axetil Acute sinusitis: Amoxicillin-Clavulanate, Azithromycin, Cefdinir, Cefprozil, Cefuroxime Axetil Streptococcal pharyngitis: Amoxicillin-Clavulanate, Azithromycin, Cefadroxil, Cefdinir, Cefprozil, Cefuroxime Axetil, Cephalexin
- Total: Total of all reporting groups
Arm/Group | Narrow Spectrum Antibiotics | Non-narrow Spectrum Antibiotics | Total
Number analyzed (Participants) | 1604 | 868 | 2472
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4.83 (3.51) | 5.19 (3.56) | 4.96 (3.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 774 | 423 | 1197
  Male | 830 | 445 | 1275
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Latino/hispanic | 147 | 65 | 212
  Race/Ethnicity: White (non-latino or unknown ethnicity) | 821 | 630 | 1451
  Race/Ethnicity: Black (non-latino or unknown ethnicity) | 474 | 106 | 580
  Race/Ethnicity: Other (non-latino/unknown ethnicity) | 129 | 59 | 188
  Race/Ethnicity: Unknown race and unknown ethnicity | 33 | 8 | 41
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1604 | 868 | 2472

OUTCOME MEASURES:

1. Primary Outcome: Health Related Quality of Life Score
Description: The health related quality of life score was obtained using the PedsQL(TM) (Mapi Research Trust, Lyon, France. www.pedsql.org) Parent-Proxy Report Generic Core Scales and Parent Report Infant Scales administered during the 5-10 day interview. Briefly, the PedsQL(TM) is a 23-item questionnaire assessing developmentally appropriate metrics (questions vary by age group: 1-12 months, 13-24 months, 2-4 years, 5-7 years, 8-12 years) related to core dimensions of health and role functioning. Our primary outcome was the Total Scale Score, which is a summary score of physical, emotional, social, and school functioning. The score range is zero to 100 and higher scores indicate a better health-related quality of life.
Time Frame: 5-10 days after ARTI diagnosis
Population: 1 subject did not respond to enough of the questions to obtain a score; 41 children missing race and ethnicity were excluded
Measure: Geometric Mean (Standard Deviation); unit: scores on a scale
Groups:
- Broad Spectrum Antibiotic: Children diagnosed with an ARTI and prescribed a broad spectrum antibiotic
Arm/Group | Narrow Spectrum Antibiotic | Broad Spectrum Antibiotic
Number analyzed (Participants) | 1570 | 860
scores on a scale | 91.5 (9.3) | 90.2 (10.5)
Statistical Analysis 1: Comparison: Narrow Spectrum Antibiotic vs Broad Spectrum Antibiotic; Propensity-score based full matching performed using patient and physician-level characteristics. Average treatment effect weights calculated and applied to a weighted linear regression; Test type: Superiority or Other; p = 0.008, Weighted linear regression; Propensity-score based full matching performed. Average treatment effect weights calculated and applied to a weighted linear regression; Score difference = -1.40, 95% CI 2-sided [-2.44 to -0.36] — Narrow antibiotics is the reference group. A score difference less than zero indicates that broad spectrum antibiotics are associated with a lower (poorer) health related quality of life score

2. Secondary Outcome: Missed School or Daycare From Illness
Description: Among children who attend school or daycare, child had to miss school or day care due to illness
Time Frame: 5-10 days after ARTI diagnosis
Population: Among children who attend school or daycare; 41 children missing race and ethnicity were excluded
Measure: Count of Participants; unit: Participants
Arm/Group | Narrow Spectrum Antibiotic | Broad Spectrum Antibiotic
Number analyzed (Participants) | 1199 | 702
Participants | 503 | 305
Statistical Analysis 1: Comparison: Narrow Spectrum Antibiotic vs Broad Spectrum Antibiotic; Propensity-score based full matching performed using patient and physician-level characteristics. Average treatment effect weights calculated and applied to a weighted logistic regression. Risk difference obtained by marginal standardization; Test type: Superiority or Other; p = 0.39, Weighted logistic regression; Propensity-score based full matching. Average treatment effect weights calculated and applied to a weighted logistic regression; Risk Difference (RD) = 2.4, 95% CI 2-sided [-3.1 to 7.9] — Broad spectrum antibiotics are the reference. A risk difference more than 0 indicates that the broad spectrum antibiotics had a higher risk of adverse outcome

3. Secondary Outcome: Required Additional Childcare
Description: Among children who attend school or daycare, parent or another caretaker had to miss work or an obligation due to child's illness OR additional childcare had to be sought for the child.
Time Frame: 5-10 days after ARTI diagnosis
Population: Among children who attend school or daycare; 41 children missing race and ethnicity were excluded
Measure: Count of Participants; unit: Participants
Groups:
- Non-narrow Spectrum Antibiotic: Children diagnosed with an ARTI and prescribed a non-narrow spectrum antibiotic
Arm/Group | Narrow Spectrum Antibiotic | Non-narrow Spectrum Antibiotic
Number analyzed (Participants) | 1190 | 701
Participants | 390 | 220
Statistical Analysis 1: Comparison: Narrow Spectrum Antibiotic vs Non-narrow Spectrum Antibiotic; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.59, Weighted logistic regression; [statistical method as in outcome 2, analysis 1]; Risk Difference (RD) = 1.5, 95% CI 2-sided [-3.9 to 6.8] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Experience Side Effects
Description: Child experienced a side effect including: rash, diarrhea or upset stomach/vomiting
Time Frame: 14-20 days after ARTI diagnosis
Population: Question was asked in the 14-20 interview so some subjects were lost to follow-up; 41 children missing race and ethnicity were excluded
Measure: Count of Participants; unit: Participants
Arm/Group | Narrow Spectrum Antibiotic | Non-narrow Spectrum Antibiotic
Number analyzed (Participants) | 1360 | 725
Participants | 341 | 258
Statistical Analysis 1: Comparison: Narrow Spectrum Antibiotic vs Non-narrow Spectrum Antibiotic; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Weighted logistic regression; [statistical method as in outcome 2, analysis 1]; Risk Difference (RD) = 12.2, 95% CI 2-sided [7.3 to 17.2] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Symptoms Present on Day 3
Description: During 5-10 day interview, parents were asked about symptoms related to child's illness (otitis media: fever, ear pain, decreased appetite; sinusitis: fever, face/head pain, decreased appetite; pharyngitis: throat pain, fever, decreased appetite). Parent was asked if symptoms was present at diagnosis. If yes, had the symptom resolved. If yes, when. We assessed whether symptoms present at day 3 after diagnosis.
Time Frame: 3 days after ARTI diagnosis
Population: Among subjects who reported having at least one symptom at the time of diagnosis; 41 children missing race and ethnicity were excluded
Measure: Count of Participants; unit: Participants
Arm/Group | Narrow Spectrum Antibiotic | Non-narrow Spectrum Antibiotic
Number analyzed (Participants) | 1128 | 647
Participants | 427 | 267
Statistical Analysis 1: Comparison: Narrow Spectrum Antibiotic vs Non-narrow Spectrum Antibiotic; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.09, Weighted logistic regression; [statistical method as in outcome 2, analysis 1]; Risk Difference (RD) = 4.9, 95% CI 2-sided [-0.8 to 10.6] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Sleep Disturbance
Description: The PedsQL questionnaire includes one or two questions, depending on age, about sleep. For children <24 months, parents are asked the frequency (never, almost never, sometimes, often, almost always) their child has (1) "difficulty falling asleep" and (2) "difficulty sleeping through the night." For children ≥2 years, parents are asked the frequency their child has "trouble sleeping." We categorized children as either without sleep disturbance ("Never" for each sleep question) or with sleep disturbance. Outcome measure shows the number of participants with sleep disturbance.
Time Frame: Days 5-10 Interview
Population: 41 children missing race and ethnicity excluded; 1 child did not complete PedsQL
Measure: Count of Participants; unit: Participants
Arm/Group | Narrow Spectrum Antibiotic | Broad-Spectrum Antibiotic
Number analyzed (Participants) | 1570 | 860
Participants | 582 | 378
Statistical Analysis 1: Comparison: Narrow Spectrum Antibiotic vs Broad-Spectrum Antibiotic; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.07, Weighted logistic regression; [statistical method as in outcome 2, analysis 1]; Risk Difference (RD) = 4.6, 95% CI 2-sided [-0.3 to 9.6] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to 20 days from ARTI diagnosis
Description: Adverse events were assessed at the interview that occurred between day 14 and day 20 after diagnosis. Subjects with missing data due to incomplete interviews or withdrawal/loss to follow-up prior to that interview are not included. All-cause mortality and SAEs could be determined for all subjects via reviews of electronic health records.
Arm/Group | Narrow Spectrum Antibiotic | Broad Spectrum Antibiotic
All-Cause Mortality (participants affected / at risk) | 0/1604 | 0/868
Serious Adverse Events (participants affected / at risk) | 0/1604 | 0/868
Other Adverse Events (participants affected / at risk) | 345/1367 | 258/726
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Narrow Spectrum Antibiotic (N=1367) | Broad Spectrum Antibiotic (N=726)
Diarrhea (General disorders) | 216 | 203
Rash (General disorders) | 150 | 90
Upset stomach and/or vomiting (General disorders) | 80 | 50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes